CLINICAL TRIAL: NCT04968275
Title: A Randomized Pilot Trial of a Cannabis Harm Reduction e-Intervention (CHAMPS) for Young Adults With Early Psychosis Who Use Cannabis
Brief Title: A Cannabis Harm Reduction e-Intervention for Young Cannabis Users With Early Psychosis
Acronym: CHAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20.433
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Psychotic Disorder; Marijuana Use; Young Adult
Keywords: Psychosis; Cannabis; Youth
MeSH Terms: conditions — Psychotic Disorders; Marijuana Use; Marijuana Abuse | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: two-arm parallel, open-labelled, pilot randomized controlled trial
Masking Description: Group assignment will not be masked after randomization, but it will be at the data analysis stage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHAMPS and EIS (Experimental): The Cannabis Harm-reducing App for Managing Practices Safely (CHAMPS) is a brief harm reduction e-intervention based on the principles of motivational interviewing and harm reduction approaches. This e-intervention will be completed by the participant using a smart phone. There will be a total of six individual sessions each lasting 15-20 min. There will be one booster session offered at 4 weeks post-intervention to review goal setting, evaluate motivation around changing cannabis use practices. This e-intervention will be administered adjunctively to psychosis early intervention services (EIS).
  Interventions: Behavioral: CHAMPS
- EIS alone (No Intervention): Early intervention services (EIS) for psychosis will be offered as per standard of care at participating clinical sites. Theses services vary but typically include pharmacotherapy and individual and/or group psychotherapy. Any visits and services offered in the EIS arm will be considered 'usual care' and administered either through in-person clinic visits, phone calls, or video calls. Relevant service information will be collected for study purposes.

INTERVENTIONS:
Behavioral: CHAMPS — CHAMPS provides personalized feedback on participants' cannabis use behaviors and supports strategies to change such behaviors. It comprises six modules measuring the use of cannabis protective behavioural strategies, exploring the possible benefits of changing cannabis practices and setting and monitoring the reach of a SMART cannabis use goal.
  Other Names: Technology-based psychosocial intervention; Psychotherapy
  Arms: CHAMPS and EIS

SUMMARY:
Cannabis users who experienced a psychosis are particularly vulnerable to cannabis-related harms, which can include worse psychotic symptoms and more hospitalizations. Unfortunately, few psychosocial interventions exist that aim to decrease these harms. Instead, most focus on ceasing cannabis use which is rarely appealing to cannabis users. Furthermore, face-to-face psychotherapy often remains inaccessible to people with psychosis mostly due to lack of trained clinicians. Alternatives such as e-interventions have the potential to increase access to treatment and decrease clinicians' workload. Among cannabis harm reduction approaches are the protective behavioural strategies. These strategies do not encourage nor discourage cannabis use. Instead, they recommend behaviours for safer cannabis use. For example, these strategies include: 1) avoid driving a car under the influence of cannabis, 2) avoid mixing cannabis with other drugs and 3) purchase cannabis only from a trusted source. In the present pan-Canadian study, we will test the first e-intervention called CHAMPS (Cannabis Harm-reducing App for Managing Practices Safely) for cannabis harm reduction adapted for young adult cannabis users who experienced a psychosis. CHAMPS is a smartphone application that includes 17 strategies for safer cannabis use, a personalized consumption goal and a consumption journal. The goals of this study are 1) to confirm whether CHAMPS is acceptable to participants and 2) to test whether it works, notably by positively impacting participants' health and cannabis consumption habits.

DETAILED DESCRIPTION:
This multicentric, two-arm, open-labelled, pilot randomized controlled trial involves 100 young cannabis users who experienced a psychosis and are followed in an early intervention service (EIS) in Canada. Participants will be randomized in a 1:1 ratio to one of two interventions:

* CHAMPS and EIS
* EIS alone

The smartphone application CHAMPS contains six modules (each lasting 15-20 min, weeks 1 to 6) and a booster session (20 min, week 10) based on motivational interviewing and harm reduction approaches. EIS consists of standard of care and psychoeducation material on cannabis use offered in first episode psychosis clinics and administered through in-person visits and/or phone or video calls.

All participants will be assessed for a follow-up at weeks 6, 12 and 18. Data on mental health, substance use, cannabis dependence severity, cannabis-related problems, quality of life and health care service utilization will be obtained through questionnaires and medical charts.

ELIGIBILITY:
Participants must meet all following inclusion criteria:

* diagnosed with any psychotic disorder, which can include schizophrenia, schizoaffective disorder, bipolar disorder with psychotic features, delusional disorder, psychotic disorder not otherwise specified, brief psychotic disorder and substance-induced psychotic disorder;
* has been followed at an early psychosis clinic for a minimum of 3 months;
* currently using cannabis (at least one time in the past 4 weeks);
* is open to changing cannabis-related practices;
* able to provide full informed consent;
* available for the whole study duration and able to comply with study procedures;
* able to comprehend French or English.

Participants are excluded if any of these exclusion criteria is met:

* pregnancy, nursing or any medical condition that in the opinion of the psychiatrist precludes safe participation in the study or the ability to provide fully informed consent;
* any disabling, unstable or acute mental condition that in the opinion of the psychiatrist precludes safe participation in the study or the ability to provide fully informed consent;
* any legal/judicial status/issue, pending legal action, or other reasons in the opinion of the study team that might prevent completion of the study;
* presence of a substance use disorder that, in the opinion of the psychiatrist, precludes safe participation in the study (e.g., very unstable or severe substance use disorder);
* currently seeking psychological or pharmacological treatment for cannabis use disorder to cease or decrease his/her use;
* currently participating in another specific cannabis-focused intervention.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Completion rates | Week 12
  Proportions of participants completing at least the first four CHAMPS modules or with ongoing participation in EIS.
Retention rates | Week 6
  Proportions of participants retained in the trial (completing all endpoint assessments)

SECONDARY OUTCOMES:
Acceptability (CHAMPS usage data) | Weeks -2-0 (baseline) to 10
  Number of CHAMPS modules completed, time spent on each module, time elapsed between module initiation and completion, total time spent on CHAMPS
Participant satisfaction | Weeks 6 and 12
  Score on the Client Satisfaction Questionnaire-I
Numbers of participants who are referred, screened, eligible, consenting, randomized, initiating and completing the study | Weeks -4 to 18
  Trial parameters
Efficacy (use of cannabis protective behavioral strategies) | Weeks -2-0 (baseline), 6, 12 and 18
  Change between endpoint and baseline scores on the Short Form Protective Behavioral Strategies-Marijuana questionnaire.
Efficacy (motivation to change cannabis protective behavioral strategies) | Weeks -2-0 (baseline), 6, 12 and 18
  Change between endpoint and baseline scores on the Readiness-to-Change Questionnaire modified for cannabis use

OTHER OUTCOMES:
Cannabis-related problems | Weeks -2-0 (baseline), 6, 12 and 18
  Total score on the Marijuana Problems Scale
Cannabis use | Weeks -2-0 (baseline), 6, 12 and 18
  Past two weeks cannabis use according to the Timeline Follow-Back Questionnaire
Other drug use | Weeks -2-0 (baseline), 6, 12 and 18
  Past two weeks other drug use according to the Timeline Follow-Back Questionnaire
Psychotic symptoms | Weeks -2-0 (baseline), 6, 12 and 18
  Total score on the Positive and Negative Syndrome Scale
Severity of cannabis dependence | Weeks -2-0 (baseline), 6, 12 and 18
  Total score on the Severity of Dependence Scale
Social support | Weeks -2-0 (baseline)
  Total score on the Social Provisions Scale
Health service utilization | Weeks -2-0 (baseline), 6, 12 and 18
  Past month number of emergency visits and days of hospitalization confirmed by medical record abstraction
Safety (adverse events) | Weeks 6, 12 and 18
  Adverse events and severe adverse events related or not to the study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD, MSc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (5):
- Canada (5):
  - Foothills Medical Centre Early Psychosis Intervention Program, Unit 24, 1403-29 Street NW, Calgary, Alberta
  - Nova Scotia Early Psychosis Program, 3rd Floor, Abbie Lane Bldg 5909 Veterans' Memorial Lane, Halifax, Nova Scotia
  - Clinic Connec-T - Institut universitaire en santé mentale de Montréal, 7401 rue Hochelaga, Montreal, Quebec
  - Clinique JAP, Centre hospitalier de l'Université de Montréal, 1051, rue Sanguinet, Montreal, Quebec
  - Clinic Notre-Dame des Victoires - Centre de Recherche CERVO, 2601 chemin de la Canardière, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coronado-Montoya S, Abdel-Baki A, Cote J, Crockford D, Dubreucq S, Fischer B, Lachance-Touchette P, Lecomte T, L'Heureux S, Ouellet-Plamondon C, Roy MA, Tatar O, Tibbo P, Villeneuve M, Wittevrongel A, Jutras-Aswad D. Evaluation of a Cannabis Harm Reduction Intervention for People With First-Episode Psychosis: Protocol for a Pilot Multicentric Randomized Trial. JMIR Res Protoc. 2023 Dec 18;12:e53094. doi: 10.2196/53094. PMID 38109196